CLINICAL TRIAL: NCT02872077
Title: Efficacy of Auricular Acupuncture on Neonatal Abstinence Syndrome: A Randomized Controlled Trial
Brief Title: Efficacy of Auricular Acupuncture on Neonatal Abstinence Syndrome
Acronym: AA NAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#Pro00025881
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: AA for NAS
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular Acupuncture (Active Comparator): Study subjects randomized to this group will receive auricular acupuncture: the investigator will evaluate the infant using an ear point locator to determine active sites, and will place acupuncture needles in the active sites found in one ear. Acupuncture sites will be alternated every 3 days between right and left ear.
  Interventions: Other: Auricular acupuncture
- Control (No Intervention): The subjects randomized to the control group will have NO interventions, and will continue to receive routine care for NAS, pharmacologic and non-pharmacologic, per NICU protocol.

INTERVENTIONS:
Other: Auricular acupuncture
  Arms: Auricular Acupuncture

SUMMARY:
This study will assess the efficacy of needle auricular acupuncture (AA) in neonatal abstinence syndrome (NAS) infants who require pharmacologic therapy at the Tampa General Hospital NICU. The investigators will evaluate efficacy of needle AA as an adjunct treatment for NAS by means of total methadone dose exposure, peak withdrawal scores, and overall length of stay.

This is the first study to evaluate efficacy of needle AA as an adjunct treatment for NAS by means of total methadone dose exposure, peak withdrawal scores, and overall length of stay.

DETAILED DESCRIPTION:
Enrolled infants will be randomized to a control group and an acupuncture group.

The control group will receive nonpharmacologic and pharmacologic management as per our current standard of care.

The acupuncture group will additionally receive AA. Once the infant is enrolled, he/she will be randomized to the AA group or the control group. Both groups of randomized infants will be taken daily to a designated treatment room. Infants in the control group will not receive acupuncture, and will only receive observation in the treatment room and will have review of their EMR.

If in the AA group, the investigator will evaluate the infant using an ear point locator to determine active sites prior to each needle placement. Acupuncture infants will have needles placed in any active sites found in one ear (up to 5 needles). Acupuncture sites will be alternated daily between right and left ear.

Acupuncture will be discontinued on the same day as methadone is discontinued, or if infant is cleared to be discharged home on methadone, acupuncture is discontinued when infant reaches the discharge dose of methadone.

Data for both groups will be collected on the day of enrollment, every three days during study participation, and at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥ 35 0/7 weeks assessed by the obstetrical team from dating of last menstrual period, ultrasound, or best obstetric estimate
2. Admitted to the TGH Transition Nursery or NICU with a diagnosis of NAS, or maternal / infant positive urine drug screen result
3. May have any of the following additional diagnoses at the time of admission: late prematurity, hyperbilirubinemia, hypoglycemia, sepsis without hypotension, respiratory distress without requiring support, or temperature instability
4. Parents give written consent prior to starting pharmacologic treatment for NAS
5. AA needles are placed within 9 hours of infant's initial NICU Finnegan score >4

Exclusion Criteria:

1. Helix or antihelix of ear is deformed and needle is unable to be placed
2. Skin condition around the ear
3. A suspected or confirmed genetic or metabolic syndrome
4. Department of Children and Families investigation results in termination of parental rights

Max Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-08; Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
The number of infants requiring / starting methadone | Up to 5 days

SECONDARY OUTCOMES:
cumulative total amount of methadone exposure | up to two months
total length of hospital stay | duration of hospital stay
peak single finnegan score after treatment initiation | within first two weeks
Peak dose of methadone required after initial AA treatment | within the first two weeks
average modified finnegan neonatal abstinence severity score for CNS symptoms | Up to two months
  1. Excessive cry
  2. Sleep <3 hours after feeding
  3. Hyperactive reflexes
  4. Tremors
  5. Increased muscle tone
  6. Excoriation
  7. Myoclonic jerks
  8. Generalized convulsions

CONTACTS AND LOCATIONS:
Overall Officials: Maya Balakrishnan, MD, Study Director — USF Health Pediatrics / Neonatology
Locations (1):
- USF Health, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No